CLINICAL TRIAL: NCT00735371
Title: A Phase III, Randomized, Double-Blind, Multi-Center, Parallel-Group, Placebo-Controlled, Forced-dose Titration, Safety and Efficacy Study of Lisdexamfetamine Dimesylate (LDX) in Adolescents Aged 13-17 With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Efficacy and Safety of Lisdexamfetamine Dimesylate (LDX) in Adolescents With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-305
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2010-02-23 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lisdexamfetamine Dimesylate (LDX) 30 mg (Active Comparator)
  Interventions: Drug: LDX 30 mg
- LDX 50 mg (Active Comparator)
  Interventions: Drug: LDX 50 mg
- LDX 70 mg (Active Comparator)
  Interventions: Drug: LDX 70 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LDX 30 mg — Eligible subjects will be randomized in a 1:1:1:1 ratio to a daily morning dose of LDX (30, 50, or 70mg/day) or placebo for a double-blind stepwise forced dose titration (3 weeks) followed by a 1-week Dose Maintenance Period. The test product is LDX, available in 30, 50, and 70mg capsules. All test products will appear identical to placebo to protect the study blind.
  Other Names: Vyvanse
  Arms: Lisdexamfetamine Dimesylate (LDX) 30 mg
Drug: LDX 50 mg — Eligible subjects will be randomized in a 1:1:1:1 ratio to a daily morning dose of LDX (30, 50, or 70mg/day) or placebo for a double-blind stepwise forced dose titration (3 weeks) followed by a 1-week Dose Maintenance Period. The test product is LDX, available in 30, 50, and 70mg capsules. All test products will appear identical to placebo to protect the study blind.
  Arms: LDX 50 mg
Drug: LDX 70 mg — Eligible subjects will be randomized in a 1:1:1:1 ratio to a daily morning dose of LDX (30, 50, or 70mg/day) or placebo for a double-blind stepwise forced dose titration (3 weeks) followed by a 1-week Dose Maintenance Period. The test product is LDX, available in 30, 50, and 70mg capsules. All test products will appear identical to placebo to protect the study blind.
  Arms: LDX 70 mg
Drug: Placebo — Placebo will be identical to test product.
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy of LDX treatment group compared to placebo on the change from Baseline ADHD-RS-IV score at endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV-TR criteria for a primary diagnosis of ADHD
* Baseline ADHD-RS-IV score >=28
* BP w/in 95th percentile for age, gender, and height

Exclusion Criteria:

* Subject has controlled or uncontrolled comorbid psychiatric diagnosis
* Subject has conduct disorder
* Suicidal
* Under or overweight
* Concurrent chronic or acute illness that might confound results.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 314 (Actual)
Dates: Start 2008-10-08 (Actual); Primary Completion 2009-04-06 (Actual); Study Completion 2009-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (45):
- United States (45):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Valley Clinical Research, Inc., El Centro, California
  - Peninsula Research Associates, Inc, Rolling Hills Estates, California
  - Psychiatric Centers at San Diego (PCSD-Feighner Research Institute), San Diego, California
  - Elite Clinical Trials, Inc, Wildomar, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Amedica Research Institute, Inc., Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Janus Center for Psychiatric Research, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Clinco Inc., Terre Haute, Indiana
  - Cientifica, Inc at Prairie View, Newton, Kansas
  - Psychiatric Associates, Overland Park, Kansas
  - Vince and Associates Clinical Research, Inc., Overland Park, Kansas
  - Pedia Research, LLC, Owensboro, Kentucky
  - Four Rivers Clinical Research, Inc., Paducah, Kentucky
  - Louisiana Research Associates, Inc, New Orleans, Louisiana
  - Bart Sangal, MD, Troy, Michigan
  - Center for Psychiatry and Behavioral Medicine, Inc, Las Vegas, Nevada
  - Children's Specialized Hospital, Toms River, New Jersey
  - Bioscience Research, LLC, Mount Kisco, New York
  - Triangle Neuropsychiatry, PLLC, Durham, North Carolina
  - Innovis Health/Odyssey Research, Fargo, North Dakota
  - University Hospitals of Cleveland Division of Child Adolescent Psychiatry, Cleveland, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - OCCI, Eugene, Oregon
  - Summit Research Network, Portland, Oregon
  - OCCI Inc, Salem, Oregon
  - CRI Worldwide, Philadelphia, Pennsylvania
  - Youth and Family Research Program/WP IC ADHD Research Program, Pittsburgh, Pennsylvania
  - Valerie Arnold, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Bayou City Research, Ltd, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - ADHD Clinic of San Antonio, San Antonio, Texas
  - Vermont Clinical Study Center, Burlington, Vermont
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Neuroscience, Inc, Herndon, Virginia
  - Dominion Clinical Research, Midlothian, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

REFERENCES:
- [Result] Findling RL, Childress AC, Cutler AJ, Gasior M, Hamdani M, Ferreira-Cornwell MC, Squires L. Efficacy and safety of lisdexamfetamine dimesylate in adolescents with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2011 Apr;50(4):395-405. doi: 10.1016/j.jaac.2011.01.007. Epub 2011 Mar 3. PMID 21421179
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisdexamfetamine Dimesylate (LDX) 30 mg; LDX 50 mg; LDX 70 mg: Subjects will be randomized in a 1:1:1:1 ratio to a daily morning dose of Lisdexamfetamine dimesylate (LDX) 30, 50, or 70mg/day or placebo for a double-blind stepwise forced dose titration (3 weeks) followed by a 1-week Dose Maintenance Period.
- Placebo: Placebo
Period: Overall Study
Arm/Group | Lisdexamfetamine Dimesylate (LDX) 30 mg | LDX 50 mg | LDX 70 mg | Placebo
Started | 78 | 79 | 78 | 79
Completed | 63 | 66 | 67 | 69
Not Completed | 15 | 13 | 11 | 10
Not completed — Adverse Event | 3 | 3 | 4 | 1
Not completed — Protocol Violation | 2 | 2 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 3 | 1
Not completed — Lack of Efficacy | 4 | 2 | 0 | 4
Not completed — Sponsor Decision | 3 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 2 | 0
Not completed — Prior Vyvanse Exposure | 1 | 1 | 0 | 0
Not completed — Exclusion criteria | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine Dimesylate (LDX) 30 mg | LDX 50 mg | LDX 70 mg | Placebo | Total
Number analyzed (Participants) | 78 | 79 | 78 | 79 | 314
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 78 | 79 | 78 | 79 | 314
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.39) | 14.7 (1.29) | 14.4 (1.30) | 14.5 (1.25) | 14.6 (1.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 34 | 25 | 94
  Male | 59 | 63 | 44 | 54 | 220
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78 | 79 | 78 | 79 | 314

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale-fourth Edition (ADHD-RS-IV) Total Score at up to 4 Weeks
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and 1, 2, 3 and 4 weeks
Population: Full Analysis Set (FAS) is defined as all subjects who took at least one dose of study medication and had a valid Baseline and at least one post-Baseline follow-up assessment of the primary outcome measure (ADHD-RS-IV Total Score)
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) 30 mg | LDX 50 mg | LDX 70 mg | Placebo
Number analyzed (Participants) | 78 | 76 | 78 | 77
Units on a scale | -18.3 (1.25) | -21.1 (1.28) | -20.7 (1.25) | -12.8 (1.25)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) 30 mg vs Placebo; Test type: Superiority or Other; p = 0.0056, ANCOVA
Statistical Analysis 2: Comparison: LDX 50 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: LDX 70 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: Number of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) Scores
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 1, 2, 3 and 4 Weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX) 30 mg | LDX 50 mg | LDX 70 mg | Placebo
Number analyzed (Participants) | 78 | 76 | 78 | 77
Participants | 44 | 53 | 57 | 30
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate (LDX) 30 mg vs Placebo; Test type: Superiority or Other; p = 0.0235, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: LDX 50 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: LDX 70 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Youth Quality of Life-Research Version (YQOL-R) Total Score
Description: The Youth Quality of Life-research version (YQOL-R) is a validated 56-item generic instrument for comparing quality of life of adolescents across condition groups that scores each question on a scale from 0 (never) to 4 (very often). The YQOL scores are transformed to a 0-100 scale for easy interpretability. Higher scores indicate better quality of life.
Time Frame: Baseline and 4 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lisdexamfetamine Dimesylate (LDX) 30 mg | LDX 50 mg | LDX 70 mg | Placebo
Number analyzed (Participants) | 78 | 76 | 78 | 77
Units on a scale
  Baseline | 79.3 (10.03) | 80.5 (10.63) | 78.8 (15.38) | 79.2 (11.08)
  4 Weeks | 81.1 (11.09) | 81.3 (11.86) | 81.3 (14.66) | 81.3 (12.16)

ADVERSE EVENTS:
Description: Safety Population defined as all subjects who took at least one dose of study medication.
Arm/Group | Lisdexamfetamine Dimesylate (LDX) 30 mg | LDX 50 mg | LDX 70 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/77 | 0/78 | 0/77
Other Adverse Events (participants affected / at risk) | 51/78 | 53/77 | 56/78 | 38/77
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lisdexamfetamine Dimesylate (LDX) 30 mg (N=78) | LDX 50 mg (N=77) | LDX 70 mg (N=78) | Placebo (N=77)
Decreased appetite (Metabolism and nutrition disorders) | 29 | 21 | 29 | 2
Headache (Nervous system disorders) | 9 | 13 | 12 | 10
Insomnia (Psychiatric disorders) | 7 | 8 | 11 | 3
Weight decreased (Investigations) | 3 | 7 | 12 | 0
Irritability (General disorders) | 6 | 2 | 8 | 3
Fatigue (General disorders) | 4 | 2 | 4 | 2
Dizziness (Nervous system disorders) | 1 | 4 | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 4 | 4 | 6
Nausea (Gastrointestinal disorders) | 1 | 3 | 5 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 6 | 4 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.